CLINICAL TRIAL: NCT05190796
Title: Relationship Between Platelet Indices and Recurrent Pregnancy Loss
Brief Title: Platelet Indices and Recurrent Pregnancy Loss
Status: Completed | Type: Observational
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohamed Elsibai Anter, Assistant professor of obstetrics and gynecology, Menoufia University
Other Study IDs: 19819OBSGN26
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Abortion, Recurrent
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women with history of recurrent pregnancy loss.: 100 women who had history of recurrent pregnancy loss.
  Interventions: Other: platelet indices
- women without history of recurrent pregnancy loss.: 50 women who had given birth at term (>37 weeks of gestation) to healthy infants (control group)
  Interventions: Other: platelet indices

INTERVENTIONS:
Other: platelet indices — One sample of 20 mL venous blood was drawn by standard phlebotomy from all of the participants. This sample was kept for the evaluation of hemoglobin, hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW), erythrocyte count, leukocyte count, platelet count, platelet distribution width (PDW), MPV and plateletcrit by means of an automated commercial counter (Coulter counter, Max Instruments Laboratory). After this venous blood sample was conveyed into a sodium citrate tube, it was transported in a temperature-controlled container and collected in plastic provettes (Falcon blue cap) containing 3 mL of 3.8% sodium citrate dihydrate and 136 mM glucosium. Then the samples were sent to the laboratory.

SUMMARY:
The aim of this study was to evaluate relationship between platelet indices, red blood cell indices and recurrent pregnancy loss.

DETAILED DESCRIPTION:
Recurrent pregnancy loss is defined as three or more consecutive pregnancy losses at or less than 20 weeks of gestation or with a fetal weight less than 500 gram. The American society for reproductive medicine (2008) proposed that recurrent pregnancy loss is defined as two or more failed clinical pregnancies confirmed by either sonographic or histopathological examination.The etiology of recurrent pregnancy loss is multifactorial and include uterine anomalies, endocrinological disorders, immunological causes, infection, chromosomal abnormalities and maternal autoimmune diseases. However, the underlying cause cannot be clarified in 50-60% of all recurrent pregnancy miscarriages.Accumulating evidence supports the concept that abnormalities of blood coagulation, generically defined as the presence of a prothrombotic state (congenital or acquired), plays an important role in adverse pregnancy outcome and is the basis of 40-70% of cases of recurrent abortions or unexplained sterility. In addition to development of many pregnancy complications such as preeclampsia, intrauterine growth restriction, preterm labor, preterm pre-labor rupture of membranes and fetal demise, recognize the same mechanism .Pregnancy causes many alterations in hemostatic balance that leading to a tendency towards thrombophilia. Such a tendency is considered as a mechanism that compensates for the hemostatic challenge of delivery. Thrombophilia in pregnancy is due to the increase in several clotting factors, including factor I, factor VII, factor VIII and von Willebrand. Moreover other markers reflecting hypercoagulability (such as D-dimer and/or prothrombin fragment) are increased during pregnancy .Red cell distribution width is a red cell parameter that measures the variability of red cell volume/size (anisocytosis). Red cell distribution width can be reported statistically as RDW-CV (coefficient of variation) or RDW-SD (standard deviation). RDW-SD is an actual measurement of the width of the erythrocyte distribution curve (measured at a relative height of 20% above the baseline).Reference range: 39-46fL .RDW-CV is calculated from standard deviation and MCV. RDW-CV: 1SD/MCV x 100, reference Range: 11.6-14.6% (Cholada and Eris, 2015), (Curry and Staros, 2015). 11.6-14.6% platelet distribution width is an indicator of variation in the size of platelet which may be a sign of activation of platelets. PDW is a simple, practical and more specific marker of platelet activation. An increased PDW is an indication for the anisocytosis of platelets. Standard PDW ranges from 9 to 14 fL (Aynioglu et al., 2014).

ELIGIBILITY:
Inclusion Criteria:

* patients with Recurrent miscarriage is defined as three or more consecutive pregnancy losses at or less than 20 weeks of gestation or with a fetal weight less than 500 grams

Exclusion Criteria:

* A woman who had experienced recurrent pregnancy loss due to uterine anomalies, diabetes mellitus and thyroid disease.
* Hypertensive women.
* Patients with coagulation defects.
* History of deep vein thrombosis or pulmonary thromboembolism.
* Use of medications affecting platelet functions such as aspirin, nonsteroidal anti-inflammatory drugs, oral contraceptives, hormonal treatments, anti-platelet, and anticoagulant drugs.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: This study included 150 subjects attending outpatient clinic of menoufia university hospital and were divided into two groups:
  * Group A: 100 women who had history of recurrent pregnancy loss.
  * Group B: 50 women who had given birth at term (>37 weeks of gestation) to healthy infants (control group).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Mean Platelet Volume | 1 day
  a measure of the average size of the platelet, expressed in femtolitre (fL)
plateletcrit (PCT) | 1 day
  a measure of total platelet mass, expressed in percentage (%)
Platelet Distribution Width (PDW) | 1 day
  a measure that reflects variation of platelet size distribution, expressed in femtolitre (fL)

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University hospital, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No